CLINICAL TRIAL: NCT01565863
Title: The Progressive Goal Attainment Program for Veterans Project
Brief Title: Progressive Goal Attainment Program for Veterans
Acronym: PGAP for Vets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); The Boeing Company (Industry); Bristol-Myers Squibb (Industry); The Community Foundation for Greater New Haven (Unknown); Disabled American Veterans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PGAP for Vets 1166.01.410.10
Record Dates: First submitted 2012-03-23; First posted 2012-03-29 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Mental Disorders; Worries; Pain or Disability
Keywords: Perceived Disability; Mental Wellness; Employment; Social Integration and Engagement; Goal Achievement
MeSH Terms: conditions — Mental Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Goal Attainment Program (Experimental)
  Interventions: Behavioral: Progressive Goal Attainment Program
- VA employment services (No Intervention)

INTERVENTIONS:
Behavioral: Progressive Goal Attainment Program — The Progressive Goal Attainment Program (PGAP) is a behavioral intervention originally developed in Canada at McGill University in order to increase return to work and community integration for individuals who receive worker's compensation. PGAP is the first disability program that is specifically designed to target the psycho-social risk factors of disability. The premise behind PGAP is that inactivity and attitudinal barriers increase work disability, and these issues are a primary cause of unemployment for individuals with physical and mental disabilities. PGAP is a structured, 10-week intervention that focuses upon helping clients develop a planned activity schedule to assist them in resuming desirable life activities.
  Other Names: PGAP
  Arms: Progressive Goal Attainment Program

SUMMARY:
The purpose of this study is to test the effectiveness of the Progressive Goal Attainment Program (PGAP) in improving employment outcomes and community engagement among U.S. veterans with disabilities.

DETAILED DESCRIPTION:
Veterans with disabilities often have low self-esteem and motivation, significant depression and a belief that their disability precludes them from gainful employment. The Progressive Goal Attainment Program (PGAP) is specifically designed to target these psycho-social risk factors of disability. PGAP is a structured, 10-week intervention that focuses on helping clients develop a planned activity schedule to assist them in resuming desirable life activities, including employment. The PGAP for Veterans Project will test the feasibility of delivering PGAP to U.S. military veterans. The research will focus on the best means of service delivery, staffing needs and how to coordinate PGAP in a larger veteran service system. MDRC will also gather information on the target population, recruitment methods, the feasibility of scaling and replication, and employment outcomes among the sample. Two hundred veterans will be enrolled and randomly assigned into the study across two sites: Errera Community Care Center within (part of the VA Connecticut Health Care System) and the Michael DeBakey VA Medical Center in Houston, Texas.

ELIGIBILITY:
Inclusion Criteria:

* Self-reporting a disability.
* Unemployed or under-employed.
* Likely to benefit from PGAP (i.e. unengaged in social and community activities, difficulty attaining work due to motivational factors).

Exclusion Criteria:

* Does not consent to be in the study.
* Significant barriers: serious substance abuse, significant psychotic disorders and cognitive disabilities that would preclude them from active participation in PGAP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Employment | 6 months

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Lehman Quality of Life Interview: Participants to rate their level of satisfaction with several domains of their lives (e.g. daily activities, social relations etc.) and their feelings about their lives as a whole on a 1-7 ("delighted" to "terrible") scale.
Citizenship | 6 months
  Citizenship Measure: 42-item scale that asks about the person's involvement in community and social activities and their ability to act and make choices on their own behalf on a 1-5 ("not at all/never" to "a lot/very often") scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Baird, Study Director — MDRC; Jack Tsai, Principal Investigator — VA Connecticut Healthcare System; Anthony Kerrigan, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (2):
- United States (2):
  - VA Connecticut Health Care Center, West Haven, Connecticut
  - Michael E. DeBakey VA Medical Center, Houston, Texas

REFERENCES:
- [Background] Adams H, Ellis T, Stanish WD, Sullivan MJ. Psychosocial factors related to return to work following rehabilitation of whiplash injuries. J Occup Rehabil. 2007 Jun;17(2):305-15. doi: 10.1007/s10926-007-9082-3. Epub 2007 May 8. PMID 17486435
- [Background] Sullivan MJ, Adams H, Rhodenizer T, Stanish WD. A psychosocial risk factor--targeted intervention for the prevention of chronic pain and disability following whiplash injury. Phys Ther. 2006 Jan;86(1):8-18. doi: 10.1093/ptj/86.1.8. PMID 16386058
- [Background] Sullivan MJ, Feuerstein M, Gatchel R, Linton SJ, Pransky G. Integrating psychosocial and behavioral interventions to achieve optimal rehabilitation outcomes. J Occup Rehabil. 2005 Dec;15(4):475-89. doi: 10.1007/s10926-005-8029-9. PMID 16254750
- [Background] Hossain F, Baird P, and Pardoe R. Improving employment outcomes and community integration for veterans with disabilities: Early implementation of the Progressive Goal Attainment Program (PGAP) for Veterans Demonstration. April 2013. New York: MDRC.
- See also: The Progressive Goal Attainment Program (PGAP) — http://www.pdp-pgap.com/pgap/en/index.html
- See also: Link to working paper with results cited above — http://www.mdrc.org/publication/improving-employment-outcomes-and-community-integration-veterans-disabilities